CLINICAL TRIAL: NCT00154726
Title: A Phase II Study of Weekly Paclitaxel(Taxol)and 24-Hour Infusion High-Dose 5-Fluorouracil and Leucovorin(HDFL)in the Treatment Locally Advanced and Recurrent/Metastatic Gastric Cancers
Brief Title: Paclitaxel-HDFL for Locally Advanced and Recurrent/Metastatic Gastric Cancers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 36-3
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2005-11-22 (Estimated); Status verified 2005-08

CONDITIONS: Locally Advanced and Recurrent/Metastatic Gastric Cancer
Keywords: Paclitaxel-HDFL,Locally Advanced and Recurrent/Metastatic Gastric Cancer
MeSH Terms: conditions — Recurrence; Stomach Neoplasms

INTERVENTIONS:
Drug: Paclitaxel-HDFL

SUMMARY:
The purpose of this study is to evaluate the efficacy,response rate,time to treatment failure,overall survival,toxicities of Paclitaxel-HDFL regimen in locally advanced/inoperable and recurrent/metastatic gastric cancers. To evaluate the resectability and relapse pattern after potentially curative resection of neoadjuvant Paclitaxel-HDFL regimen

DETAILED DESCRIPTION:
In the treatment of metastatic breast cancer, paclitaxel followed by weekly HDFL has been shown to have a 55% response rate in anthracycline-resistant patient. Recently, regimen combining paclitaxel and moderately-high-dose 5-FU (1500mg/m2) has had response rate up to 61.5% (including 23%CR) in a small group of gastric cancer patients (8 responders in 13 patients). Thus, the sequential use of weekly paclitaxel followed by weekly HDFL regimen may become a new generation of chemotherapeutic regimen for the treatment of gastric cancer. Further study with a larger group of patients and further testing of possible schedules of administration are warranted.

ELIGIBILITY:
Inclusion Criteria: 1.Histologically or cytologically confirmed gastric adenocarcinoma 2.Measurable or evaluable disease 3.No previous C/T 4.Age 18 ~ 70 years 5.KPS >=60% 6.WBC>=4,000, pltate>=100K, Creatinine<=1.5mg/dl, serum bil<=1x UNL, transaminase<=3.5x ULN

Exclusion Criteria: 1.CNS metastasis 2.Patients receive concomitant anti-cancer C/T or R/T 3.Patients who are pregnant and with an expected life expectancy less than 3months 4.Symptomatic heart disease,active infection, extensive liver disease or liver cirrhosis 5.TG<=70mg/dl 6.Mental status is not fit for clinical trial

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 1997-04; Study Completion 2005-08

PRIMARY OUTCOMES:
Response rate

SECONDARY OUTCOMES:
overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Ann-Lii Cheng, M.D.,Ph.D., Study Chair — Department of Oncology, National Taiwan University Hospital